CLINICAL TRIAL: NCT04714749
Title: Feasibility and Tolerance Study for the Treatment of Varicose Ulcers by Cyanoacrylate Glue
Brief Title: Feasibility and Tolerance Study for the Treatment of Varicose Ulcers by Cyanoacrylate Glue (ETUVVE)
Acronym: ETUVVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Pasteur (Other)
Responsible Party: Principal Investigator, Nicolas NEAUME, Principal investigator, MD, Clinique Pasteur
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A02799-30
Record Dates: First submitted 2021-01-13; First posted 2021-01-19 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Venous Leg Ulcer
Keywords: endovenous treatment; glue
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endovenous treatment (Experimental): Endovenous treatment with cyanoacrylate glue
  Interventions: Procedure: Endovenous treatment; Device: Cyanoacrylate glue

INTERVENTIONS:
Procedure: Endovenous treatment — Treatment of great saphenous vein (its tributaries and possible incompetent perforators feeding the ulcer) by endovascular cyanoacrylate glue
Device: Cyanoacrylate glue — Treatment of great saphenous vein (its tributaries and possible incompetent perforators feeding the ulcer) by endovascular cyanoacrylate glue

SUMMARY:
Ulcers of the lower limbs are a major public health problem whose management needs to be further improved, particularly in terms of healing time, prevalence and recurrence rate. Ulcers of venous origin, or mixed arteriovenous and predominantly venous, represent the majority of leg ulcers with an estimated proportion of 70 to 80% of cases. These are painful, disabling conditions that are difficult to treat in a lasting way.

This study focuses on a treatment strategy with endovascular glue. The advantage of treating ulcers with cyanoacrylate glue is the possibility of occluding the great saphenous vein over its entire length, freeing itself from neurological complications secondary to endovenous thermal techniques (laser, radiofrequency), as well as the possibility of treating by direct puncture any perforators or tributaries feeding the ulcer.

This treatment strategy would improve the healing process for a lasting resolution of this pathology. This study aims to describe the feasibility and tolerance of this type of treatment in the resolution of varicose ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Primary insufficiency of the great saphenous vein (GVS) by a reflux> 0.5 second from the inter-fascial saphenous trunk to the upper 1/3 of the thigh extending over the entire height of the thigh either in the saphenous compartment or in at least one extra-fascial tributary, in a standing patient, by compression of the calf
* CEAP: C6, ulcer present on a single leg whose size can be captured by a simple photograph
* Diameter of the GVS at the saphenofemoral junction ≥3 or ≤12 millimeters
* Patient affiliated or beneficiary of a social security scheme
* Patient having signed the informed consent

Exclusion Criteria:

* Patient with a circumferential ulcer
* Patient with ipsilateral small saphenous vein insufficiency
* Presenting a serious current pathology and / or a life expectancy of less than 5 years
* History of deep or superficial vein thrombosis in the previous 6 months
* Patient with arteriopathy obliterating of the affected lower limb, with an IPS <0.8 or> 1.3
* With post-thrombotic obstructive syndrome in the popliteal and / or femoral and / or iliac stage on the ipsilateral lower limb
* Presenting primary or post-thrombotic axial deep venous reflux on the ipsilateral lower limb
* Suspicion of non-post-thrombotic iliac compression on Doppler ultrasound
* Contraindication to the intended treatment technique
* Known allergy to cyanoacrylate glue or xylocaine
* Patient with a BMI greater than 40 (morbid obesity)
* Patient whose geographical distance is not compatible with the follow-up of the study
* Pregnant or breastfeeding woman
* Patient participating in another clinical study
* Patient linguistically or psychically unable to understand the information given, to give informed consent or to answer the study questionnaires.
* Protected patients: Adults under some guardianship or other legal protection; Hospitalized without consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Ulcer healing | Between surgery and 12 months after
  Proportion of patients who presented with healing of the venous ulcer

SECONDARY OUTCOMES:
Functional and technical success | Day 0, Day 8, Month 1, Month 6 , Month 12
  Success assessed by occlusion of treated veins
VAS Pain | Day 0, Day 8, Month 1, Month 6 , Month 12
  Visual analogue scale (0-100 mm); higher is worse
Severity | Day 0, Day 8, Month 1, Month 6 , Month 12
  Clinical Venous Severity Score (CVSS); score between 0 to 30; higher is worse
Healing | Between surgery and 12 months after
  Time to ulcer healing
Ulcer duration | Between surgery and 12 months after
  Time without ulcer; time to recurrence (in days )
Ulcer recurrence | Between surgery and 12 months after
  Rate of recurrence
Symptoms | Day 0, Day 8, Month 1, Month 6 , Month 12
  VEINES Sym (VEnous INsufficiency Epidemiologic and Economic Study - Symptoms) questionnaire
Patient Quality of Life | Day 0, Day 8, Month 1, Month 6 , Month 12
  VEINES QOL (VEnous INsufficiency Epidemiologic and Economic Study- Quality Of Life) Questionnaire
Adverse events | Day 0, Day 8, Month 1, Month 6 , Month 12
  Adverse events related to glue or to the endovenous intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas NEAUME, MD, Principal Investigator — Clinique Pasteur
Locations (1):
- Clinique Pasteur Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gohel MS, Barwell JR, Taylor M, Chant T, Foy C, Earnshaw JJ, Heather BP, Mitchell DC, Whyman MR, Poskitt KR. Long term results of compression therapy alone versus compression plus surgery in chronic venous ulceration (ESCHAR): randomised controlled trial. BMJ. 2007 Jul 14;335(7610):83. doi: 10.1136/bmj.39216.542442.BE. Epub 2007 Jun 1. PMID 17545185
- [Background] Gohel MS, Heatley F, Liu X, Bradbury A, Bulbulia R, Cullum N, Epstein DM, Nyamekye I, Poskitt KR, Renton S, Warwick J, Davies AH; EVRA Trial Investigators. A Randomized Trial of Early Endovenous Ablation in Venous Ulceration. N Engl J Med. 2018 May 31;378(22):2105-2114. doi: 10.1056/NEJMoa1801214. Epub 2018 Apr 24. PMID 29688123
- [Background] Hirsch T. Varicose vein therapy and nerve lesions. Vasa. 2017 Mar;46(2):96-100. doi: 10.1024/0301-1526/a000588. Epub 2016 Dec 16. PMID 27981883
- [Background] Toonder IM, Lam YL, Lawson J, Wittens CH. Cyanoacrylate adhesive perforator embolization (CAPE) of incompetent perforating veins of the leg, a feasibility study. Phlebology. 2014 May;29(1 suppl):49-54. doi: 10.1177/0268355514529696. Epub 2014 May 19. PMID 24843086
- [Background] Morrison N, Gibson K, Vasquez M, Weiss R, Jones A. Five-year extension study of patients from a randomized clinical trial (VeClose) comparing cyanoacrylate closure versus radiofrequency ablation for the treatment of incompetent great saphenous veins. J Vasc Surg Venous Lymphat Disord. 2020 Nov;8(6):978-989. doi: 10.1016/j.jvsv.2019.12.080. Epub 2020 Mar 20. PMID 32205125
- [Background] Heatley F, Onida S, Davies AH. The global management of leg ulceration: Pre early venous reflux ablation trial. Phlebology. 2020 Sep;35(8):576-582. doi: 10.1177/0268355520917847. Epub 2020 Apr 8. PMID 32268842
- [Background] Abenhaim L, Kurz X. The VEINES study (VEnous Insufficiency Epidemiologic and Economic Study): an international cohort study on chronic venous disorders of the leg. VEINES Group. Angiology. 1997 Jan;48(1):59-66. doi: 10.1177/000331979704800110. PMID 8995345
- [Background] Lamping DL, Schroter S, Kurz X, Kahn SR, Abenhaim L. Evaluation of outcomes in chronic venous disorders of the leg: development of a scientifically rigorous, patient-reported measure of symptoms and quality of life. J Vasc Surg. 2003 Feb;37(2):410-9. doi: 10.1067/mva.2003.152. PMID 12563215
- [Background] Kahn SR, Lamping DL, Ducruet T, Arsenault L, Miron MJ, Roussin A, Desmarais S, Joyal F, Kassis J, Solymoss S, Desjardins L, Johri M, Shrier I; VETO Study investigators. VEINES-QOL/Sym questionnaire was a reliable and valid disease-specific quality of life measure for deep venous thrombosis. J Clin Epidemiol. 2006 Oct;59(10):1049-56. doi: 10.1016/j.jclinepi.2005.10.016. Epub 2006 Jun 23. PMID 16980144
- [Background] Bland JM, Dumville JC, Ashby RL, Gabe R, Stubbs N, Adderley U, Kang'ombe AR, Cullum NA. Validation of the VEINES-QOL quality of life instrument in venous leg ulcers: repeatability and validity study embedded in a randomised clinical trial. BMC Cardiovasc Disord. 2015 Aug 11;15:85. doi: 10.1186/s12872-015-0080-7. PMID 26260973